CLINICAL TRIAL: NCT00057187
Title: Improving Substance Abuse Treatment Aftercare Adherence and Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Virginia Polytechnic Institute and State University (Other); Duke University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 99-282
Record Dates: First submitted 2003-03-27; First posted 2003-03-31 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Substance Dependence; Compliance; Treatment Outcome
MeSH Terms: conditions — Substance-Related Disorders; Patient Compliance | interventions — Contracts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Contracting, Prompting and Reinforcing

INTERVENTIONS:
Behavioral: Contracting, Prompting and Reinforcing

SUMMARY:
Although substance abuse treatment continuing care participation is strongly related to positive treatment outcomes, participation rates are low and few interventions have been developed that improve continuing care adherence and outcome.

DETAILED DESCRIPTION:
Background:

Although substance abuse treatment continuing care participation is strongly related to positive treatment outcomes, participation rates are low and few interventions have been developed that improve continuing care adherence and outcome.

Objectives:

The objectives of the study were: 1) to compare the effectiveness of an aftercare intervention consisting of a participation contract, attendance prompts, and attendance reinforcers (CPR) to a standard treatment (STX) on adherence to therapy; and 2) to assess the effects of this intervention on treatment outcome

Methods:

We recruited 150 veterans from the Salem VAMC�s SARRTP who could participate in aftercare. Our population is similar to those in other VA�s (97% male, 54% Caucasian, 46% minority, 49 years mean age, 44% alcohol dependent only, 56% drug dependent, and 44% with a dual diagnosis). In this randomized clinical trial, treatment adherence and outcome were measured at baseline and 3-, 6- and 12-months after participants entered treatment using interviews, questionnaires, alcohol and drug screens, VA medical records, and therapist ratings. The study design is a repeated measures nested cohort design, with an intervention and a standard care group. The primary outcome, abstinence rate, will be analyzed using a logistic regression model in which the parameters of interest are estimated using Generalized Estimating Equations (GEE).

Status:

Participant recruitment and follow-up interviews were completed in June 2003 and August 2004, respectively. The HSR&D final report was submitted in April 2005. The main results paper and additional papers will be submitted for publication in 2005.

ELIGIBILITY:
Inclusion Criteria:

All graduates of the Salem VA's SARRTP who: live within a 60 minute drive of the Salem VAMC, or 1 of our 5 SARRTP outreach clinics; have transportation and a job schedule that allows them to attend outpatient aftercare therapy.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Lash, PhD, Principal Investigator — Salem VA Medical Center, Salem, VA
Locations (1):
- Salem VA Medical Center, Salem, VA, Salem, Virginia, United States

REFERENCES:
- [Result] Lash SJ, Burden JL, Monteleone BR, Lehmann LP. Social reinforcement of substance abuse treatment aftercare participation: Impact on outcome. Addict Behav. 2004 Feb;29(2):337-42. doi: 10.1016/j.addbeh.2003.08.008. PMID 14732421
- [Result] DeMarce JM, Lash SJ, Stephens RS, Grambow SC, Burden JL. Promoting continuing care adherence among substance abusers with co-occurring psychiatric disorders following residential treatment. Addict Behav. 2008 Sep;33(9):1104-12. doi: 10.1016/j.addbeh.2008.02.008. Epub 2008 Feb 23. PMID 18573617
- [Result] DeMarce JM, Burden JL, Lash SJ, Stephens RS, Grambow SC. Convergent validity of the Timeline Followback for persons with comorbid psychiatric disorders engaged in residential substance use treatment. Addict Behav. 2007 Aug;32(8):1582-92. doi: 10.1016/j.addbeh.2006.11.015. Epub 2007 Jan 24. PMID 17254716
- [Result] Lash J, Burden L, Fearer A. Contracting, Prompting and Reinforcing Substance Abuse Treatment Aftercare Adherence. Journal of Drug Addiction, Education and Eradication. 2007 Jul 1; 2(3/4):455-490.
- [Result] Lash SJ, Stephens RS, Burden JL, Grambow SC, DeMarce JM, Jones ME, Lozano BE, Jeffreys AS, Fearer SA, Horner RD. Contracting, prompting, and reinforcing substance use disorder continuing care: a randomized clinical trial. Psychol Addict Behav. 2007 Sep;21(3):387-97. doi: 10.1037/0893-164X.21.3.387. PMID 17874889